CLINICAL TRIAL: NCT05066932
Title: Advanced Lipoproptein Profiling and Cardiovascular Risk Stratification in Familial Hypercholesterolemia
Acronym: CARDIOMET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210455; 2021-A00747-34 (Other: ANSM)
Record Dates: First submitted 2021-09-09; First posted 2021-10-04 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-01

CONDITIONS: Familial Hypercholesterolemia; Atherosclerosis
Keywords: Familial hypercholesterolemia; Primary prevention; Apolipoproteins; Atherosclerosis
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Familial Hypercholesterolemia and hyperTriglyceridemia: Patients with Familial Hypercholesterolemia and hyperTriglyceridemia
  Interventions: Other: Additionnal blood samples
- Familial Hypercholesterolemia without hyperTriglyceridemia: Patients with Familial Hypercholesterolemia and without hyperTriglyceridemia
  Interventions: Other: Additionnal blood samples

INTERVENTIONS:
Other: Additionnal blood samples — Additionnal blood samples

SUMMARY:
Familial hypercholesterolaemia (FH) is a genetic disorder characterised by elevated plasma LDLC levels.

The causal role of low-density lipoprotein cholesterol (LDLC) in the progression of cardiovascular disease (CVD) is indisputable: genetic, epidemiological and interventional trials have unanimously shown that a reduction in LDL-C is associated with a reduced risk of CVD.

Some drawbacks related to the limitations of the analytical methods are slowly surfacing due to the lower LDLC target achieved with the combination of several new treatments. This is mainly due to the fact that LDLC is not a comprehensive marker to stratify cardiovascular risk in subjects with increased levels of other atherogenic lipoproteins.

Direct measurement of the concentration of apolipoproteins involved in cholesterol and triglycerides transportation, may provide more information than the simple measure of the cholesterol contained in these particles. There is an interest in measuring the various players involved in the lipoprotein processing chain. These apolipoproteins are increasingly being considered as possible biomarkers of cardiovascular disease risk.

Indeed, there is increasing evidence that advanced lipoprotein testing methods, such as multiplexed measurements of apolipoprotein panels (ApoA-I, A-II, A-IV, B-100, C-I, C-II, C-III, E), provide more detailed information on the dyslipidaemic profiles of patients compared to conventional lipid testing, finally allowing a better understanding and stratification of subclinical atherosclerosis in these patients.

The main objective of this study is to compare the apolipoprotein profile of patients with FH by comparing those with associated hypertriglyceridemia (hyperTG) to those with isolated hypercholesterolaemia.

Adult subjects with a molecular diagnosis of Familial Hypercholesterolemia, treated by a statin, on primary prevention, asymptomatic for cardiovascular symptoms, will be recruited and stratified according to the presence/absence of hyperTG in a case-control prospective observational study design.

DETAILED DESCRIPTION:
The crucial role of dyslipidaemia, in particular hypercholesterolaemia, in the development of cardiovascular diseases is particularly well documented. The causal role of LDLC in the progression of CVD is indisputable: genetic, epidemiological and interventional trials have unanimously shown that a reduction in LDL-C is associated with a reduced risk of CVD.

Some drawbacks related to the limitations of the analytical methods are slowly surfacing due to the lower LDLC target achieved with the combination of several new treatments. This is mainly due to the fact that LDLC is not a comprehensive marker to stratify cardiovascular risk in subjects with increased levels of other atherogenic lipoproteins.

Familial hypercholesterolaemia (FH) is a genetic disorder characterised by elevated plasma LDLC levels.

Plasma levels of key lipoproteins, including LDLC levels, are major determinants and triggers of vascular endothelial damage; monocyte to macrophage differentiation and foam cell formation, leading to the development of atherosclerotic lesions; premature coronary artery disease (CAD); peripheral arterial disease; and supra-aortic stenosis. The earlier these events occur, the higher the cholesterol level.

A growing body of experimental and clinical evidence suggests that triglyceride-rich lipoproteins (TRL), and in particular remnant particles, contribute to atherogenesis and thus to the progression of cardiovascular disease.

In addition, these lipids such as cholesterol and triglycerides (TG) circulate in blood plasma as lipoproteins, supramolecular assemblies whose structure is provided by specific proteins: apolipoproteins.

Direct measurement of the concentration of atherogenic particles involved in the metabolism of cholesterol and TG could therefore provide more information than simply measuring the cholesterol contained in these particles. There is an interest in measuring the various players involved in the lipoprotein processing chain. These apolipoproteins are increasingly being considered as possible biomarkers of cardiovascular disease risk. Indeed, there is increasing evidence that advanced lipoprotein testing methods, such as multiplexed measurements of apolipoprotein panels (ApoA-I, A-II, A-IV, B-100, C-I, C-II, C-III, E), provide more detailed information on the dyslipidaemic profiles of patients compared to conventional lipid testing, allowing for a better understanding and stratification of subclinical atherosclerosis in these patients.

Primary objective:

To compare the apolipoprotein profile of patients with FH by comparing those with associated hyperTG to those with isolated hypercholesterolaemia.

Secondary objectives:

Compare the subclinical impairment of FH patients with and without hyperTG

* Compare the coronary atherosclerotic burden, assessed by the Calcium Score
* Compare carotid atherosclerotic burden, assessed by echodoppler
* Compare femoral atherosclerotic burden, assessed by echodoppler

Conduct of the research :

The patient will be informed of the study and if agree to participate, additional blood tubes will be collected for the research during the blood sampling carried out as part of the usual care.

Analysis will be performed in collaboration with LNE, the France's national metrology laboratory as part of the European CARDIOMET project.

A biobank and serum library will also be constituted during the study for further and additional analysis.

Two groups of patients will be enrolled :

* patients with familial hypercholesterolaemia (FH) and hypertriglyceridemia (hyperTG)
* patients with familial hypercholesterolaemia (FH) without hypertriglyceridemia (hyperTG)

ELIGIBILITY:
Inclusion Criteria:

A. Patients with familial hypercholesterolemia (FH) and with hyperTG :

1. Age > 18 years
2. Molecular or clinical diagnosis of FH
3. Primary prevention (no coronary artery disease, cerebrovascular disease or lower limb arterial disease)
4. HyperTG or TG levels between 135-500 mg/dl on statin therapy
5. Patient informed of the research, not having objected to participation and having provided written consent for genetic analysis

B. Patients with familial hypercholesterolemia (FH) and without hyperTG :

1. Age > 18 years
2. Mild diagnosis
3. Primary prevention (no coronary artery disease, cerebrovascular disease or lower limb arterial disease)
4. TG <135mg/dl on statin therapy
5. Patient informed of the research, did not object to participation and provided written consent for genetic testing

Exclusion Criteria:

1. Secondary prevention or planned coronary intervention or cardiac surgery
2. History of acute or chronic pancreatitis
3. Statin-intolerant patient
4. Glycated haemoglobin level greater than 10.0%.
5. Human Immunodeficiency Virus infection on treatment,
6. Use of corticosteroids
7. Severe renal impairment (Glomerular filtration rate < 30 ml/min)
8. Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with familial hypercholesterolemia (FH), with or without hyperTG
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Apolipoprotein score | At day 1
  Apolipoprotein score (ApoA-I, A-II, A-IV, B-100, C-I, C-II, C-III, E) will be measured in gram per liter (g/l) and assessed by liquid chromatography-mass spectrometry (LC-MS).

SECONDARY OUTCOMES:
Calcium score | At day 1
  The Calcium score will be measured in Hounsfield units (HU) and assessed using the Agatston method (such examination will be performed as part of the usual management of care).
Intima-media thickening of the distal common carotid artery | At day 1
  Measurement of intima-media thickening of the distal common carotid artery, quantified by Doppler ultrasound using semi-automated calculation software.
Presence of carotid plaque | At day 1
  Presence of carotid plaque assessed by the European Carotid Surgery Trial (ECST) method
Intima-media thickening of the distal common femoral artery | At day 1
  Measurement of intima-media thickening of the distal common femoral artery, quantified by Doppler ultrasound using semi-automated calculation software.
Presence of femoral plaque | At day 1
  Presence of femoral plaque assessed by the European Carotid Surgery Trial (ECST) method

CONTACTS AND LOCATIONS:
Overall Officials: Eric BRUCKERT, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital de la Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided